CLINICAL TRIAL: NCT06206967
Title: Rehabilitation Program for Promotion Active Lifestyle After Suffering a Pulmonary Thromboembolism
Brief Title: Promotion of Active Lifestyle in Thromboembolism Patients
Acronym: ACTIVATEP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Marie Carmen Valenza, UNIVERSITY PROFESSOR, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DF0099UG
Record Dates: First submitted 2023-11-15; First posted 2024-01-16 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Pulmonary Thromboembolism
Keywords: Pulmonary Thromboembolism; Rehabilitation; Activity Promotion
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Activity Promotion Group (Experimental): The rehabilitation program has the purpose of motivating patients to be more physically active. The treatment protocol had a total duration of 12 weeks.
  Three sessions are conducted during hospitalization for the education of patients and to start physical activity. A diary is provided to patients to record the activities that they perform during each week until completing the 12 weeks.
  Additionally, phone calls are performed at 15 days, 1 and 2 months to motivate patients and answer any questions they may have.
  Interventions: Other: Physical Activity Promotion
- Control group (Active Comparator): Patients received an informational brochure in a consultation with a health professional. The brochure explained the importance of physical activity to improve the health condition of these patients. Patients had the opportunity to ask any questions to the healthcare professional.
  Interventions: Other: Control Intervention

INTERVENTIONS:
Other: Physical Activity Promotion — This intervention includes a hospital-based and a home-based intervention. During the hospital stay, the patients were provided with a health education which included information about thromboembolism pathophysiology and its management, healthy-lifestyle habits, benefits of early-mobilisation, and any questions patients may have would be answered.
  Additionally, an early-mobilization program is provided, which includes resistance and aerobic exercise.
  At the end of the hospital stay, a diary is provided to patients for recording the physical activity that performing the following 3 months. This diary is accompanied by phone calls at 15 days, 1 and 2 months of the hospital stay. During the phone calls, patients are motivated to increase their activity levels, and any questions patients may have, are answered.
  Other Names: Motivation for being more physically active
  Arms: Physical Activity Promotion Group
Other: Control Intervention — Patients received an informational brochure in a consultation with a health professional. The brochure explained the importance of physical activity to improve the health condition of these patients. Patients had the opportunity to ask any questions to the healthcare professional.
  Arms: Control group

SUMMARY:
Patients who have suffered a pulmonary thromboembolism used to reduce their activity levels because of the symptoms and the fear to suffer other pulmonary thromboembolism. These patients often have sequelae after the hospitalization that previous studies have associated with a lack of physical activity.

The main objective of this research is to investigate the efficacy of a rehabilitation program for promotion higher activity levels in quality of life and self-perceived discapacity of thromboembolism patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes.
* Agreed to participate.
* Thromboembolism patients meeting the diagnosis criteria for this disease.

Exclusion Criteria:

* Neurological or orthopaedic pathologies that limited voluntary movement.
* Cognitive impairment that prevented them from understanding and answering the questionnaires.
* Patients suffering from a previous pulmonary thromboembolism.
* Patients who don´t understand Spanish language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-01-20 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Changes in discapacity | Baseline
  Changes in self-perceived discapacity were measured using the World Health Organization Disability Assessment Schedule, WHODAS 2.0, which provides a global measure of disability and 7 domain-specific scores.
Changes in discapacity | Immediately after the hospital stay
  Changes in self-perceived discapacity were measured using the World Health Organization Disability Assessment Schedule, WHODAS 2.0, which provides a global measure of disability and 7 domain-specific scores. The punctuation range from 36 to 144, and higher score indicate higher disability, worse.
Changes in discapacity | At 12 weeks at the hospital discharge
  Changes in self-perceived discapacity were measured using the World Health Organization Disability Assessment Schedule, WHODAS 2.0, which provides a global measure of disability and 7 domain-specific scores. The punctuation range from 36 to 144, and higher score indicate higher disability, worse.
Quality of life measure with EuroQol-5D-5L | Baseline
  Changes in quality of life were measured using the Euroqol 5dimensions which comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. It also includes a visual analogue scale to report the health status from 0 to 100.
Quality of life measure with EuroQol-5D-5L | Immediately after the hospital stay
  Changes in quality of life were measured using the Euroqol 5dimensions which comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. It also includes a visual analogue scale to report the health status from 0 to 100.
Quality of life measure with EuroQol-5D-5L | At 12 weeks at the hospital discharge
  Changes in quality of life were measured using the Euroqol 5dimensions which comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. It also includes a visual analogue scale to report the health status from 0 to 100.
Physical Activity Levels measured wit IPAQ | Baseline
  The International Physical Activity Questionnaire (IPAQ) was developed to measure health-related physical activity (PA) in populations. The activities are classified as vigorous, moderate and walking, and total METs are calculated. NO minimum or maximum valors are stablished. Higher scores indicates higher physical activity levels. Better.
Physical Activity Levels measured wit IPAQ | At 12 weeks at the hospital discharge
  The International Physical Activity Questionnaire (IPAQ) was developed to measure health-related physical activity (PA) in populations. The activities are classified as vigorous, moderate and walking, and total METs are calculated. NO minimum or maximum valors are stablished. Higher scores indicates higher physical activity levels. Better.

SECONDARY OUTCOMES:
Dyspnoea | Baseline
  The perceived dyspnoea is measure with the Borg Scale. This scale in range from 0-10, where higher score indicate higher levels of dyspnoea. Worse.
Dyspnoea | Immediately after the hospital stay
  The perceived dyspnoea is measure with the Borg Scale. This scale in range from 0-10, where higher score indicate higher levels of dyspnoea. Worse.
Dyspnoea | At 12 weeks at the hospital discharge
  The perceived dyspnoea is measure with the Borg Scale. This scale in range from 0-10, where higher score indicate higher levels of dyspnoea. Worse.
Changes in Psycho-emotional status | Baseline
  The DASS-21 scale asks respondents to answer 21 questions focused on experiencing symptoms of depression, anxiety, and stress in the past week.
  Participants were provided four response options: 0=never, 1=sometimes, 2=a lot of the time, 3=most or all of the time. Higher response values, and higher scores, indicate higher levels of experiencing the condition measured.
Changes in Psycho-emotional status | Hospital Discharge
  The DASS-21 scale asks respondents to answer 21 questions focused on experiencing symptoms of depression, anxiety, and stress in the past week.
  Participants were provided four response options: 0=never, 1=sometimes, 2=a lot of the time, 3=most or all of the time. Higher response values, and higher scores, indicate higher levels of experiencing the condition measured.
Changes in Psycho-emotional status | At 12 weeks at the hospital discharge
  The DASS-21 scale asks respondents to answer 21 questions focused on experiencing symptoms of depression, anxiety, and stress in the past week.
  Participants were provided four response options: 0=never, 1=sometimes, 2=a lot of the time, 3=most or all of the time. Higher response values, and higher scores, indicate higher levels of experiencing the condition measured.
Changes in Performance status | Baseline
  The performance status is measure with the Canadian Occupational Performance Measure. In a semi structured interview, the patient is encouraged to discuss areas of activity that may present problems that they may need to, want to, or are expected to carry out on a regular basis. These problem areas are then rated in terms of importance to the patient´s life using the rating scale from 1 - 10, where 1 = not at all important, and 10 = extremely important to the client. The five most important problems are then the focus of intervention and the outcome measurement. The patient, using a similar scale, is then asked to rate his/her perception of performance and satisfaction with this performance in the selected problem areas. The two scores are separately summed and divided by the number of problem areas, giving the mean foreach.
Changes in Performance status | Immediately after the hospital stay
  The performance status is measure with the Canadian Occupational Performance Measure. In a semi structured interview, the patient is encouraged to discuss areas of activity that may present problems that they may need to, want to, or are expected to carry out on a regular basis. These problem areas are then rated in terms of importance to the patient´s life using the rating scale from 1 - 10, where 1 = not at all important, and 10 = extremely important to the client. The five most important problems are then the focus of intervention and the outcome measurement. The patient, using a similar scale, is then asked to rate his/her perception of performance and satisfaction with this performance in the selected problem areas. The two scores are separately summed and divided by the number of problem areas, giving the mean foreach.
Changes in Performance status | At 12 weeks at the hospital discharge
  The performance status is measure with the Canadian Occupational Performance Measure. In a semi structured interview, the patient is encouraged to discuss areas of activity that may present problems that they may need to, want to, or are expected to carry out on a regular basis. These problem areas are then rated in terms of importance to the patient´s life using the rating scale from 1 - 10, where 1 = not at all important, and 10 = extremely important to the client. The five most important problems are then the focus of intervention and the outcome measurement. The patient, using a similar scale, is then asked to rate his/her perception of performance and satisfaction with this performance in the selected problem areas. The two scores are separately summed and divided by the number of problem areas, giving the mean foreach.
Changes in Breathlessness Beliefs | Baseline
  The Breathlessness Beliefs Questionnaire (BBQ) is a concise 10-item self-report assessment tool used in the realm of respiratory health. It gauges an individual's perceptions and beliefs regarding breathlessness or dyspnea. Respondents rate their agreement with statements on a scale, often ranging from 0 to 10, reflecting their thoughts about the causes, consequences, and controllability of breathlessness. Higher scores may indicate more negative beliefs, while lower scores suggest more positive or adaptive beliefs. The BBQ aids in tailoring interventions and treatments for individuals with respiratory conditions, shedding light on the cognitive factors contributing to breathlessness-related distress and ultimately improving patient well-being and functional outcomes.
Changes in Breathlessness Beliefs | Immediately after the hospital stay
  The Breathlessness Beliefs Questionnaire (BBQ) is a concise 10-item self-report assessment tool used in the realm of respiratory health. It gauges an individual's perceptions and beliefs regarding breathlessness or dyspnea. Respondents rate their agreement with statements on a scale, often ranging from 0 to 10, reflecting their thoughts about the causes, consequences, and controllability of breathlessness. Higher scores may indicate more negative beliefs, while lower scores suggest more positive or adaptive beliefs. The BBQ aids in tailoring interventions and treatments for individuals with respiratory conditions, shedding light on the cognitive factors contributing to breathlessness-related distress and ultimately improving patient well-being and functional outcomes.
Changes in Breathlessness Beliefs | At 12 weeks at the hospital discharge
  The Breathlessness Beliefs Questionnaire (BBQ) is a concise 10-item self-report assessment tool used in the realm of respiratory health. It gauges an individual's perceptions and beliefs regarding breathlessness or dyspnea. Respondents rate their agreement with statements on a scale, often ranging from 0 to 10, reflecting their thoughts about the causes, consequences, and controllability of breathlessness. Higher scores may indicate more negative beliefs, while lower scores suggest more positive or adaptive beliefs. The BBQ aids in tailoring interventions and treatments for individuals with respiratory conditions, shedding light on the cognitive factors contributing to breathlessness-related distress and ultimately improving patient well-being and functional outcomes.
Changes in managing the own healthcare | Immediately after the hospital stay
  The Patient Activation Measure-13 (PAM-13) is a concise assessment tool designed to evaluate an individual's knowledge, skills, and confidence in managing their own healthcare. Comprising 13 items, this self-report questionnaire helps healthcare professionals and researchers gauge a patient's level of activation and engagement in their healthcare journey. Respondents answer a series of questions related to their health-related knowledge, confidence in managing their health, and their proactivity in seeking healthcare information and making informed decisions. Higher PAM-13 scores indicate a higher level of patient activation, which is often associated with better health outcomes and more effective self-management of chronic conditions. This tool plays a crucial role in tailoring patient education and support strategies.
Changes in managing the own healthcare | At 12 weeks at the hospital discharge
  The Patient Activation Measure-13 (PAM-13) is a concise assessment tool designed to evaluate an individual's knowledge, skills, and confidence in managing their own healthcare. Comprising 13 items, this self-report questionnaire helps healthcare professionals and researchers gauge a patient's level of activation and engagement in their healthcare journey. Respondents answer a series of questions related to their health-related knowledge, confidence in managing their health, and their proactivity in seeking healthcare information and making informed decisions. Higher PAM-13 scores indicate a higher level of patient activation, which is often associated with better health outcomes and more effective self-management of chronic conditions. This tool plays a crucial role in tailoring patient education and support strategies.
Changes in physical functioning | Baseline
  The physical functioning is measured using the "Short Physical Performance Battery" (SPPB). To assess usual walking speed (meters/second), the participants were asked to walk 4 metro at their regular pace twice from a standing position. The standing balance tests included side-by-side, semi-tandem, and full-tandem standing, and the participants were timed until they moved, or 10 s had elapsed. To assess the 5-times sit-to-stand test, the participants were asked to perform five chair stands as quickly as possible. Time (in seconds) was registered with a stopwatch with a resolution of 0.01 s. The total score ranged from 0 (worst) to 12 points (best). An increase of 1-point is recommended in disability research.
Changes in physical functioning | Immediately after the hospital stay
  The physical functioning is measured using the "Short Physical Performance Battery" (SPPB). To assess usual walking speed (meters/second), the participants were asked to walk 4 metro at their regular pace twice from a standing position. The standing balance tests included side-by-side, semi-tandem, and full-tandem standing, and the participants were timed until they moved, or 10 s had elapsed. To assess the 5-times sit-to-stand test, the participants were asked to perform five chair stands as quickly as possible. Time (in seconds) was registered with a stopwatch with a resolution of 0.01 s. The total score ranged from 0 (worst) to 12 points (best). An increase of 1-point is recommended in disability research.
Changes in physical functioning | At 12 weeks at the hospital discharge
  The physical functioning is measured using the "Short Physical Performance Battery" (SPPB). To assess usual walking speed (meters/second), the participants were asked to walk 4 metro at their regular pace twice from a standing position. The standing balance tests included side-by-side, semi-tandem, and full-tandem standing, and the participants were timed until they moved, or 10 s had elapsed. To assess the 5-times sit-to-stand test, the participants were asked to perform five chair stands as quickly as possible. Time (in seconds) was registered with a stopwatch with a resolution of 0.01 s. The total score ranged from 0 (worst) to 12 points (best). An increase of 1-point is recommended in disability research.
Changes in Maximal Grip Strength | Baseline
  Maximal grip strength was assessed using a Jamar hydraulic hand dynamometer. The participant was told to squeeze it as hard as possible and then release. This procedure was repeated three times with each hand alternating between both hands with 5 minutes rest between the trials. The grip strength was recorded in kg and the highest of the three trials was used.
Changes in Maximal Grip Strength | Immediately after the hospital stay
  Maximal grip strength was assessed using a Jamar hydraulic hand dynamometer. The participant was told to squeeze it as hard as possible and then release. This procedure was repeated three times with each hand alternating between both hands with 5 minutes rest between the trials. The grip strength was recorded in kg and the highest of the three trials was used.
Changes in Maximal Grip Strength | At 12 weeks at the hospital discharge
  Maximal grip strength was assessed using a Jamar hydraulic hand dynamometer. The participant was told to squeeze it as hard as possible and then release. This procedure was repeated three times with each hand alternating between both hands with 5 minutes rest between the trials. The grip strength was recorded in kg and the highest of the three trials was used.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Carmen Valenza, PhD, Principal Investigator — Universidad de Granada
Locations (1):
- Faculty of Health Sciences, University of Granada, Granada, Spain